CLINICAL TRIAL: NCT06490887
Title: Spine Unit Modelling Coupled With hIgh Throughput Analysis (SUIT): Targeting Degeneration With Cell Secretome
Brief Title: Spine Unit Modelling Coupled With hIgh Throughput Analysis (SUIT)
Acronym: SUIT
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: SUIT
Record Dates: First submitted 2024-03-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Disc Disease
Keywords: inflammation; degeneration; spine unit; intervertebral disc; mesenchymal stem cell
MeSH Terms: conditions — Intervertebral Disc Degeneration; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood. Collection of nucleous pulposus, annulus fibrosus and cartilaginous endplate biopsies that would be considered as waste material after surgery.
  Collection of adipose tissue that would be considered as waste material after surgery.
  Collection of amnion of human term placenta (38-40 weeks of gestation) within 6 hours of birth.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Degenerative Disc Disease patients undergoing spine surgery: Collection of blood. Collection of nucleous pulposus, annulus fibrosus and cartilaginous endplate biopsies that would be considered as waste material after surgery.
  Interventions: Other: Use of patient-derived biological samples
- Subjects undergoing plastic surgery: Collection of adipose tissue that would be considered as waste material after surgery.
  Interventions: Other: Use of patient-derived biological samples
- Pregnant female subjects: Collection of amnion of human term placenta (38-40 weeks of gestation) within 6 hours of birth.
  Interventions: Other: Use of patient-derived biological samples

INTERVENTIONS:
Other: Use of patient-derived biological samples — We will use biological samples that are routinely collected as waste material from patients undergoing surgery or from pregnant women giving birth. Peripheral blood will be also collected from patients to conduct virological screening and isolate peripheral blood mononuclear cells.

SUMMARY:
Ageing and inflammation represent two main drivers of DDD, a progressive, chronic condition involving vertebral bone, cartilaginous endplate and intervertebral disc.

In vitro investigation of the DDD-associated processes on single compartments of the spine unit or ex vivo animal models fail in recapitulating the complex spine pathophysiology or suffer from inter-species differences. Given these premises, a human organotypic model of the spine unit would represent a suitable tool to investigate the DDD-related pathways and to screen promising treatments such as MSC-based therapies.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the response of an inflamed organotypic spine unit model, intended as a 3D in vitro representation of an in vivo environment, to the treatment with mesenchymal stem cells (MSC)-derived secretome. In particular to investigate the ability of MSC-derived secretome to modulate genes found to be upregulated or downregulated by the inflammatory stimulation in the spine unit model and bring their expression back to a basal state.

Secondary aims of the study are:

* To identify specific degenerative features related to ageing and inflammation in patients affected by Degenerative Disc Disease (DDD) correlating circulating features and tissue degeneration
* To develop an organotypic spine unit model using patient-derived cells to investigate the response of cells derived from nucleus pulposus (NP), annulus fibrosus (AF) and cartilaginous endplate (CEP) to inflammation

ELIGIBILITY:
DDD patients:

* Signature of the Informed Consent for the study
* Age 30-60 years (included)
* Pfirrmann grade III-V
* Need to undergo spinal surgery

Subjects for the isolation of adipose-derived MSCs:

* Signature of the Informed Consent for the study
* Age 18-50 (included)
* Need to undergo surgery that involves the removal of adipose tissue

Subjects for the isolation of placenta-derived MSCs:

* Signature of the Informed Consent for the study
* Age 18-50 (included)
* Women who are pregnant or who have not given birth from more than 6 hours

All enrolled subjects:

- Presence of HIV, HBV, HCV or TP infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Samples will be collected from Degenerative Disc Disease patients undergoing spine surgery, from patients subjected to surgeries that involve the removal of adipose tissue and from pregnant women within 6 hours from giving birth.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of MSC-derived secretome | 30 months
  Changes in gene expression in response to the treatment of the spine unit model with MSC-derived secretome. If the MSC-derived secretome is effective, genes upregulated or downregulated by inflammatory stimulation are expected to go back to their basal levels when the inflamed model is treated with MSC-derived secretome.

SECONDARY OUTCOMES:
Characterization of patient-specific degenerative features | 30 months
  Identification of circulating degenerative features related to ageing and inflammation in patients affected by Degenerative Disc Disease (DDD) correlating with tissue degeneration.
Development of an organotypic spine unit model | 30 months
  Determination of success or failure in the development of spine unit models for each enrolled patient from which cell isolation has been successful.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, MI
  - IStituto MEditerraneo per i Trapianti e Terapie ad alta specializzazione, Palermo

IPD SHARING:
Plan to Share IPD: No